CLINICAL TRIAL: NCT05645835
Title: Dynamic Neural Systems Underlying Social-emotional Functions in Older Adults
Acronym: Dynamo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-37461; R00AG065457 (NIH); K99AG065457 (NIH)
Record Dates: First submitted 2022-11-28; First posted 2022-12-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Loneliness; Older Adults; fMRI; Emotions; EEG; Digital Intervention; Meditation
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention (Experimental): Participants will engage with the digital meditation app delivering the intervention 15 min a day, five days, a week for 6 weeks.
  Interventions: Behavioral: intervention
- waitlist control (Active Comparator): Participants will be randomized to a waitlist group for six weeks. The waitlist control group will then be able to use the meditation app for six weeks as the primary intervention group
  Interventions: Behavioral: waitlist control
- Baseline physiology (Other): A subset of participants will not participate in the intervention. Only baseline fMRI and EEG data will be collected in these participants.
  Interventions: Other: No Interventions

INTERVENTIONS:
Behavioral: intervention — the digital meditation app will be installed on participants iPad or android. Lonely older adults will use the app five days a week for six weeks total. Neuroimaging will be performed before and after the intervention.
  Arms: intervention
Behavioral: waitlist control — Participants in the waitlist group will have to wait six weeks after being screened before being able to use the meditation app after the assessment of primary and secondary endpoints
  Arms: waitlist control
Other: No Interventions — No intervention. Only baseline fMRI and EEG assessment.
  Arms: Baseline physiology

SUMMARY:
Assess the impact of a remote, app-delivered digital meditation intervention on emotional well-being of lonely older adults. Neuroimaging, electrophysiological (EEG), and autonomic physiology will be used to assess the neural correlates of the intervention. EEG and autonomic physiology will be collected while participants watch 30 min of an awe-inspiring movie. fMRI and autonomic physiology will be collected in the context of a social exploration/exploitation task.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* English language fluency
* Naive to meditation practices (not actively meditating more than one hour per month and/or meditation practice for less than a year in their entire life-time)
* No MRI contra-indications
* Cognitively healthy (no diagnosis of dementia, stroke, developmental disorders, or major systemic diseases that may impact cognitive function)

Exclusion Criteria:

* Below 60 years of age
* Not fluent in English
* Active meditator (meditating more than one hour per month and/or meditation practice for more than a year in their entire life-time).
* Presence of a severe psychiatric (e.g. schizophrenia, bipolar disorder, PTSD), neurological (epilepsy, traumatic brain injury, dementia, multiple sclerosis), or developmental disorder (e.g. autism)
* Systemic disease (e.g. major recent surgeries, cancer)
* Claustrophobia
* Contraindications for MR safety (e.g. metal in body, cochlea implants)

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in the WHO-5 Well-Being Index | Change in well-being from baseline to directly after completing the intervention (6 weeks)
  WHO-5 ranges from 0-25, with higher values indicating higher well-being

SECONDARY OUTCOMES:
Change in the 20-item UCLA loneliness scale | Change in loneliness from baseline to directly after completing the intervention (6 weeks)
  This scale ranges from 20-80, with higher values indicating higher loneliness
Change in the General Anxiety Disorder-7 (GAD-7) | Change in anxiety from baseline to directly after completing the intervention (6 weeks)
  This scale ranges from 0-21, with higher values indicating higher anxiety
Change in Psychological Stress Measure (PSM-9) | Change in stress from baseline to directly after completing the intervention (6 weeks)
  This scale ranges from 9-72, with higher values indicating higher stress
Change in Patient Health Questionnaire (PHQ-9) | Change in depression from baseline to directly after completing the intervention (6 weeks)
  This scale ranges from 0-27, with higher values indicating higher depression

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Pasquini, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No